<u>Title:</u> FES-Rowing: Preventing the Secondary Conditions of Paralysis Through Vigorous exercise-A Survey Study of User Needs

NCT Number: NCT05144113

Document Date: 06/25/2024

## **Statistical Analysis Plan**

## Data analysis

Intrapersonal (health and beliefs/attitudes) and interpersonal (friends and family) domain scores from the Barriers to Physical Activity Questionnaire for People With Mobility Impairments (BPAQ-MI) were calculated using weighted sums of the corresponding survey items. A factor correlation matrix was used to determine each item weight. Each participant's domain scores were then calculated by summing the products of each item score (0, not a barrier at all to 5, largest barrier) with each item's weight. For the Barriers to Physical Activity and Disability Survey (BPAD-S), the number of endorsements ("yes") for 19 items on distinct barriers to physical activity was counted. Participant characteristics that informed user and design needs and potential market for the at-home FES-row system were defined as the clinical diagnosis causing paralysis and type of wheelchair primarily used (i.e., manual vs. power chair). For the FES-row training group only, each participant's total score on the Quebec User Evaluation of Satisfaction With Assistive Technology (QUEST 2.0) was calculated by summing the item scores (0, least satisfied to 5, most satisfied) and dividing the sum by the number of valid responses (invalid responses were outside 0-5 range and included: "not applicable"). Data are expressed as group (FES-row and non FES-row) mean ± standard error or number (percentage of group total).

## Statistics

Between-group comparisons of demographics and questionnaire data were evaluated with two-sample t-tests when appropriate. Statistical significance will be considered at p < 0.05.

## References

1. Vasudevan, V., Rimmer, J.H., & Kviz, F. (2015). Development of the Barriers to Physical Activity Questionnaire for People with Mobility Impairments. *Disability and Health Journal*, *8*, 547-556.